CLINICAL TRIAL: NCT06020820
Title: Effectiveness Of Cervical Rehabilitation Program After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah IU Tayyaba sultan
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Post-Thyroidectomy Hypoparathyroidism
Keywords: range of motion; disability; post-thyroidectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Rehabilitation program (Intervention Group) Group A (Experimental): Positional release technique on trapezius muscle, Suboccipital muscle release, Stretching of pectoralis muscle
  Interventions: Other: Cervical Rehabilitation program (Intervention Group) Group A
- (control group) Group B (Active Comparator): neck and shoulder ROMS
  Interventions: Other: control group group B

INTERVENTIONS:
Other: Cervical Rehabilitation program (Intervention Group) Group A — (Positional release technique on trapezius muscle): the therapist locate and apply pressure along the tender points in the upper fibers of the trapezius. Lateral flexion of subject's head toward the side of a tender point held for 90 seconds.
  (Suboccipital muscle release): The therapist places both his palms under the sub occipital region of the subject with his curled-up fingers and places an upward pressure causing a stretch and distraction for 30 seconds,This technique was performed 3 times in one session.
  Stretching of pectoralis muscle:
  Pectoralis muscle stretch were performed once daily, completing three repetitions on each side with a 30-second hold. Stretching with repetition of five, three times a day for 1week neck and soulder ROMs
  Arms: Cervical Rehabilitation program (Intervention Group) Group A
Other: control group group B — 1. Relax shoulders and neck sufficiently
  2. look down
  3. turn face to the right
  4. turn face to the left
  5. incline head to the right
  6. incline head to the left
  7. turn shoulders round and round
  8. slowly raise hands fully then lower them. patients were asked to perform five repetitions of each stretching exercise, three times per day (morning, afternoon, and evening).
  Arms: (control group) Group B

SUMMARY:
The aim of this research is to determine the Effects of cervical rehabilitation program on neck pain, ROM and disability after thyroidectomy. Randomized controlled trials will be done at Pakistan ordinance factory (POF) Hospital. The sample size will be 52. The subjects were divided in two groups, with 26 subjects in Group A and 26 in Group B. Study duration was of 6 months. Sampling technique applied was Non probability Convenience Sampling technique. Both males and females of aged 30-50 years with thyroidectomy were included. Tools used in the study are Numeric Pain Rating Score (NPRS), goniometer and neck disability index (NDI).

DETAILED DESCRIPTION:
Thyroidectomy, or surgical removal of the gland, is highly recommended treatment for thyroid disorders. The most prevalent of these conditions are symptomatic benign large goiter and tumorous condition of the thyroid gland. Both younger females and postmenopausal older women are prevalent towards these disorders (nodular goiter, cancer, and hypothyroidism).

Due to hyperextended position of neck during surgery patient usually complaint about the posterior neck pain, movement difficulties of shoulder and neck, occipital headaches, shoulder stiffness, motion's cervical range of limitations and some of them experiences the discomfort symptoms such as stretching, pressing, or choking feelings in the neck, headache, shoulder stiffness, and difficulty in moving the neck or shoulders. These symptoms may persist for an extended period following surgery and may even have a negative effect on the patient's quality of life. It has been reported that hyperextension can cause bilateral hypoglossal palsy, tetraplegia and cervical artery dissection Recently, a variety of treatment modalities have been used to overcome these disturbing symptoms, such as intraoperative transcutaneous electrical nerve stimulation (TENS), preoperative bilateral greater occipital nerve (GON) block, bilateral superficial cervical plexus block combined with bilateral GON block, and postoperative neck stretching exercise. Due to surgical position of thyroidectomy patient often develops posture syndrome of thyroid surgery (PSTS), symptoms include postoperative nausea, vomiting, dizziness, headache and some discomfort associated with neck an occipital radiating pain.

Nepa Patel et al reported that both positional release technique and MET are effective for treatment of upper trapezius tightness or trigger points as the trapezius muscle works to move the neck in several directions, its degree of tightness or looseness affects neck flexibility. Om C. Wadhokar et al conducted a study on patients having neck pain with TMJ dysfunction, causes tightness of occipital muscles, difficulty in mouth opening and forward head posture. In this study suboccipital release technique was found to be more effective than conventional treatment.

In an RCT, stretching of pectoralis along with cervical mobilizations and rotation exercises were used for treatment of mechanical neck pain. And it has evaluated that it improves the active range of motion in all directions, perceived pain and disability levels. In 2019, Samah et al conducted a study to compare the effects the active neck stretching exercises and kinesio taping on patients after thyroidectomy; a significant improvement was observed in active stretching group. Another study investigated the effects of neck stretching exercises on post thyroidectomy patients with complaint of neck discomfort, and it concluded that neck stretching exercises are improving the patient disability level.

ELIGIBILITY:
Inclusion Criteria:

* • Post-thyroidectomy patients

  * Indoor patients

Exclusion Criteria:

* • Any cervical fracture/dislocations

  * Cervical instability
  * Vertebrobasilar insufficiency
  * Cervical Radiculopathy
  * Disc prolapsed at cervical region
  * Any neurological impairment

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Score (NPRS): | 1 week
  was used to assess neck pain intensity. Patients were asked to rate how bad their neck pain was on average (NPRS; range, 0, no pain, to 10, maximum pain
NDI | 1 Week
  NDI is used to asses that how neck pain affects the quality of life of a person. It consists of 10 items, from 0-5 points in each item. Total score of NDI is 50 that is converted into percentage of 100.
cervical flexion range of motion | 1 week
  the person is asked to move neck forward to touch chin and the range is taken
cervical extension range of motion | 1 week
  the person is asked to move neck backward as far as possible and the range is taken
cervical Rt rotation range of motion | 1 week
  the person is asked to move neck sideways to Rt side like saing "no" and the range is taken
cervical Lt rotation range of motion | 1 week
  the person is asked to move neck sideways to Lt side like saing "no" and the range is taken
cervical Rt side flexion range of motion | 1 week
  the person is asked to move neck sideways to Rt side like touching ear to shoulder and range is taken
cervical Lt side flexion range of motion | 1 week
  the person is asked to move neck sideways to Rt side like touching ear to shoulder and range is taken

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, Principal Investigator — Riphah International University
Locations (1):
- Pakistan ordinance factory Hospital, Wah, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No